CLINICAL TRIAL: NCT04565470
Title: Strategies of Self-management of Endometriosis Symptoms: an Observational Study
Brief Title: Strategies of Self-management of Endometriosis Symptoms
Acronym: SAGE
Status: Completed | Type: Observational
Sponsor: Benno Rehberg-Klug (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, Attending anesthesiologist, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: SAGE
Record Dates: First submitted 2020-09-19; First posted 2020-09-25 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: online questionnaire — Web-based questionnaire about use of self-management strategies

SUMMARY:
To determine the prevalence and perceived utility of self-management strategies amongst patients with endometriosis and who consult the endometriosis clinic of the Geneva University Hospital, information about these strategies will be obtained via a web-based questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients consulting at the endometriosis clinic of the HUG
* minimum 18 years
* capacity to answer the questions of the questionnaire

Exclusion Criteria:

* minor patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients consulting at a specialised centre
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
frequency of use of any self-management strategy | during the last 6 months prior to the questionnaire
  binary answer: yes/no of use

SECONDARY OUTCOMES:
frequency of use of the pre-specified strategies: gymnastics, rest, hypnosis, meditation, exercise, osteopathy, cold/warm, acupuncture, CBD, cannabis, alcohol, TENS, phytotherapy, curcuma, essential oils, diet | during the last 6 months prior to the questionnaire
  binary answer: yes/no of use

OTHER OUTCOMES:
perceived efficacy of the different strategies of self-management | during the last 6 months prior to the questionnaire
  0-10 scale for pain and 5 classes for other symptoms (none, little, medium, large, very large)
perceived reduction of analgesic use by the different strategies of self-management | during the last 6 months prior to the questionnaire
  5 classes (none, little, medium, large, very large)
side effects of the different strategies of self-management | during the last 6 months prior to the questionnaire
  free text

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rehberg-Klug, MD, Study Director — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No